CLINICAL TRIAL: NCT04311593
Title: Prognostic Value of CD Markers in Immune Thrombocytopenic Purpura
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Ahmed Mahmoud, resident doctor, Assiut University
Other Study IDs: CD markers in ITP
Record Dates: First submitted 2020-03-14; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — CD4 Lymphocyte Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: control group with normal platelet count
  Interventions: Diagnostic Test: CD4, CD19, CD38, CD56 and CD11b
- group 2: patients with acute ITP
  Interventions: Diagnostic Test: CD4, CD19, CD38, CD56 and CD11b
- group 3: patients with chronic ITP
  Interventions: Diagnostic Test: CD4, CD19, CD38, CD56 and CD11b

INTERVENTIONS:
Diagnostic Test: CD4, CD19, CD38, CD56 and CD11b — measuring CD markers by flowcytometry

SUMMARY:
In this study, we will focus on the independent prognostic relevance of the expressions of CD38, CD4, CD56, CD11b and CD19 markers in immune cells with platelet changes in patients with newly diagnosed and chronic ITP.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP), previously called idiopathic thrombocytopenia purpura, is an autoimmune disorder characterized by a severe reduction in peripheral blood platelet count. In healthy individuals, normal platelet count ranges from 150-450 × 109/L, while in thrombocytopenia counts fall to less than 100 × 109/L ( Provan et al., 2010).

Based on duration, ITP is differentiated into three phases. Newly diagnosed ITP occurs within 3 months of diagnosis, persistent ITP is present 3-12 months after diagnosis, and chronic ITP lasts >12 months since diagnosis (Roberto, 2011).

Autoantibodies against platelet glycoproteins (GPs), including GPIIb/IIIa and GPIb/IX, have been considered to play a crucial role in ITP (Nomura, 2016) . In addition to platelet destruction, impaired maturation of megakaryocytes can be associated with reduced platelet production in ITP (Muna et al., 2015).

Furthermore, considerable attention has been recently paid to the dysregulation of a new B-cell subset known as regulatory B cells (Breg) in ITP (Li et al., 2012). This B-cell subset is characterized by CD19+CD38+ expression, promoting peripheral tolerance and reducing the function of autoreactive T-helper (Th) CD4+ cells via production of interleukin 10 (IL-10) (Flores-Borja et al., 2013). So they are an interesting cell population in diseases characterized by an unbalance in the immune system, such as autoimmune diseases, chronic infections, cancer and graft rejection.( Horikawa et al., 2013).

In ITP, as a result of the defective function of Breg and also Treg (regulatory T) cells, platelet autoreactive Th CD4+ cells undergo clonal expansion (McKenzie et al., 2013). so the presence of activated platelet-specific autoreactive T cells that respond to autologous platelet antigens participating in autoantibody production in ITP via interaction with autoreactive B cells (Solanilla et al., 2005).

Since the early 1980s, many studies have documented decreased natural killer (NK) cell numbers and impairment of NK cell function in the peripheral blood of patients with autoimmune diseases such as multiple sclerosis, systemic lupus erythematosus, Sjögren's syndrome, rheumatoid arthritis, and type I diabetes (hussein et al., 2017). Furthermore, in many studies, a correlation has been found between NK cell number and activity with disease progression or remission in multiple sclerosis (MS) and systemic lupus erythematosus (SLE). (Riccieri et al., 2000).

Nk cells are identified by the expression of CD16 and CD56 surface markers, account for 5-15% of PB cells in healthy individuals .NK cells have a crucial role in the initial defense against infections in innate immunity and are particularly important in responding to viral infections (French and Yokoyama., 2004).

This finding suggests that CD16+CD56+ NK cells may play a role in the pathogenesis and prognosis of autoimmune diseases.

CD11b+ monocytes can regulate adaptive immunity by adjustment of different T-cell subsets (Kusmartsev et al., 2000). Recently showed that monocytes derived from the whole blood of chronic ITP patients promoted the development of Th CD4+ subset (Zhong et al., 2012).

Although the majority of these abnormalities can appear as the increased or decreased expressions of some CD markers in the involved cells, there have been few studies on the prognostic value of CD markers' expressions in immune cells for ITP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thrombocytopenia were identified by their medical records. According to guidelines for the investigation and management of ITP, its diagnosis in thrombocytopenic patients was based on the following criteria: the presence of thrombocytopenia (platelet counts <100 9 103/lL), patient's history, physical examination, normal concentration of hemoglobin and white blood cells (WBC), PB smear examination, normal or increased number of megakaryocytes with normal myeloid and erythroid progenitors in bone marrow (BM) smears. The absence of other diseases causing thrombocytopenia, including HIV and hepatitis C infection, SLE, aplastic anemia, megaloblastic anemia, and lymphoproliferative disorders was confirmed by BM aspiration assays. In chronic ITP : ITP patients lasting for more than 12 months

Exclusion Criteria:

* The prescence of other diseases causing thrombocytopenia, including HIV and hepatitis C infection, SLE, aplastic anemia, megaloblastic anemia and lymphoproliferative disorders was confirmed by BM aspiration assays

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Assiut university hospital - clinical hematology unit.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
measuring level of research CD markers in immue cells | one year
  in acute ITP patients : at time of diagnosis and after treatment and return of platelets count to normal count.
  in chronic ITP patients : measuring of research CD markers once.

CONTACTS AND LOCATIONS:
Overall Officials: Essam ELdeen abdmohsen mohammed, Professor, Study Director — +201001971906

REFERENCES:
- [Background] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Background] Stasi R. Pathophysiology and therapeutic options in primary immune thrombocytopenia. Blood Transfus. 2011 Jul;9(3):262-73. doi: 10.2450/2010.0080-10. Epub 2010 Nov 26. No abstract available. PMID 21251458
- [Background] Namdev R, Dutta SR, Singh H. Acute immune thrombocytopenic purpura triggered by insect bite. J Indian Soc Pedod Prev Dent. 2009 Jan-Mar;27(1):58-61. doi: 10.4103/0970-4388.50821. PMID 19414977